CLINICAL TRIAL: NCT02014272
Title: An Open Label, Single Dose, 2-Way Cross-Over Randomized Bioequivalence Study Comparing A Fixed Dose Combination Formulation, Rin 150 (Contains 150 Mg Rifampicin And 75 Mg Isoniazid Per Tablet) To An Equivalent Dose Of Single Drug Reference Preparations Of Rifampicin And Isoniazid Following Oral Administration In Healthy Adults Under Fasting Conditions
Brief Title: A Bioequivalence Study Comparing A Fixed Dose Combination Formulation, Rin 150 And Individual Reference Drugs In Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: B3801003
Record Dates: First submitted 2013-12-12; First posted 2013-12-18 (Estimated); Results first posted 2014-07-16 (Estimated); Last update posted 2014-07-16 (Estimated); Status verified 2014-06

CONDITIONS: Healthy Volunteers
Keywords: Bioequivalence; RIN 150; Healthy volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Test (Experimental): RIN 150 contains 150 rifampicin and 75 mg isoniazid
  Interventions: Drug: RIN 150
- Reference (Active Comparator): Individual references of rifampicin and isoniazid
  Interventions: Drug: reference drugs

INTERVENTIONS:
Drug: RIN 150 — Each subject will receive a single oral dose of 4 fixed dose combination tablets (RIN 150) each contains 150 rifampicin and 75 mg isoniazid.
  Arms: Test
Drug: reference drugs — Each subject will receive a single oral dose of 4 x 150 mg rifampicin capsules and 3 x 100 mg isoniazid capsules.
  Arms: Reference

SUMMARY:
This is a bioequivalence study to evaluate the bioequivalence of RIN 150 against individual reference drugs in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female, 21 to 55 years of age, body weight no less than 55 kg, with a signed and dated informed consent document and is willing and able to comply with all scheduled visits, treatment plan, laboratory tests and other study procedures.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing), positive Hepatitis B surface antigen or HIV serology results;
* Pregnant or nursing female;
* History or active tuberculosis;
* Participated in investigational drug studies within 3 months;
* Used prescription or nonprescription drugs within 7 days or 5 half-lives.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2012-09; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Singapore, Singapore, Singapore

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B3801003&StudyName=A%20Bioequivalence%20Study%20Comparing%20A%20Fixed%20Dose%20Combination%20Formulation%2C%20Rin%20150%20And%20Individual%20Reference%20Drugs%20In%20Healthy%20Volunteers

RESULTS

PARTICIPANT FLOW:
Groups:
- RIN 150 First, Then Rifampicin and Isoniazid: Single oral dose of 4 fixed dose combination (FDC) tablets of RIN 150 (each tablet contained 150 milligram [mg] rifampicin and 75 mg isoniazid) on Day 1 in first intervention period, followed by single oral dose of 4 rifampicin 150 mg capsules and 3 isoniazid 100 mg tablets on Day 1 in second intervention period. A washout period of at least 7 days was maintained between each intervention period.
- Rifampicin and Isoniazid First, Then RIN 150: Single oral dose of 4 rifampicin 150 mg capsules and 3 isoniazid 100 mg tablets on Day 1 in first intervention period followed by single oral dose of 4 fixed dose combination (FDC) tablets of RIN 150 (each tablet contains 150 mg rifampicin and 75 mg isoniazid) on Day 1 in second intervention period. A washout period of at least 7 days was maintained between each intervention period.
Period: Intervention Period 1
Arm/Group | RIN 150 First, Then Rifampicin and Isoniazid | Rifampicin and Isoniazid First, Then RIN 150
Started | 14 | 14
Completed | 13 | 13
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Adverse Event | 0 | 1
Period: Washout Period 1 (7 Days)
Arm/Group | RIN 150 First, Then Rifampicin and Isoniazid | Rifampicin and Isoniazid First, Then RIN 150
Started | 13 | 13
Completed | 13 | 13
Not Completed | 0 | 0
Period: Intervention Period 2
Arm/Group | RIN 150 First, Then Rifampicin and Isoniazid | Rifampicin and Isoniazid First, Then RIN 150
Started | 13 | 13
Completed | 13 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Analysis population included all randomized participants.
Groups:
- Entire Study Population: Includes all participants randomized to receive RIN 150 first and rifampicin and isoniazid first.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.5 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 27

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast)
Description: Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast) was reported for rifampicin and isoniazid.
Time Frame: 0 hour (pre-dose), 0.25, 0.5, 0.75, 1, 1.33 (1 hour 20 minutes), 1.67 (1 hour 40 minutes), 2, 2.33 (2 hours 20 minutes), 2.67 (2 hours 40 minutes), 3, 3.5, 4, 6, 8, 12, 16, 24 hours post-dose on Day 1
Population: Pharmacokinetic parameter analysis set included all treated participants who had at least 1 estimated pharmacokinetic parameter of primary interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (nanogram*hour) per milliliter (ng*h/mL)
Groups:
- RIN 150: Single oral dose of 4 fixed dose combination (FDC) tablets of RIN 150 (each tablet contains 150 mg rifampicin and 75 mg isoniazid) on Day 1 in either of the 2 intervention periods.
- Rifampicin and Isoniazid: Single oral dose of 4 rifampicin 150 mg capsules and 3 isoniazid 100 mg tablets on Day 1 in either of the 2 intervention periods.
Arm/Group | RIN 150 | Rifampicin and Isoniazid
Number analyzed (Participants) | 27 | 27
(nanogram*hour) per milliliter (ng*h/mL)
  AUClast: Rifampicin | 85020 (20) | 90030 (24)
  AUClast: Isoniazid | 16220 (79) | 16120 (77)
Statistical Analysis 1: Comparison: RIN 150 vs Rifampicin and Isoniazid; Natural log transformed AUClast of rifampicin was analyzed using mixed effects model with sequence,period and treatment as fixed effects and participant within sequence as random effect.The adjusted mean differences and 90% confidence intervals(CIs) for the differences were exponentiated to provide estimates of ratio of adjusted geometric means(Test/Reference) and 90% CIs for the ratios,where FDC tablet were test and single drugs were reference.Values were back-transformed from the log scale; Test type: Superiority or Other; Ratio of adjusted geometric means = 95.45, 90% CI 2-sided [92.07 to 98.94]
Statistical Analysis 2: Comparison: RIN 150 vs Rifampicin and Isoniazid; Natural log transformed AUClast of isoniazid was analyzed using mixed effects model with sequence,period and treatment as fixed effects and participant within sequence as random effect.The adjusted mean differences and 90% confidence intervals(CIs) for the differences were exponentiated to provide estimates of ratio of adjusted geometric means(Test/Reference) and 90% CIs for the ratios,where FDC tablet were test and single drugs were reference.Values were back-transformed from the log scale; Test type: Superiority or Other; Ratio of adjusted geometric means = 103.45, 90% CI 2-sided [99.33 to 107.75]

2. Primary Outcome: Maximum Observed Plasma Concentration (Cmax)
Description: Cmax was reported for rifampicin and isoniazid.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | RIN 150 | Rifampicin and Isoniazid
Number analyzed (Participants) | 27 | 27
ng/mL
  Cmax: Rifampicin | 13670 (21) | 15000 (28)
  Cmax: Isoniazid | 6080 (45) | 5577 (37)
Statistical Analysis 1: Comparison: RIN 150 vs Rifampicin and Isoniazid; Natural log transformed Cmax of rifampicin was analyzed using mixed effects model with sequence,period and treatment as fixed effects and participant within sequence as random effect.The adjusted mean differences and 90% confidence intervals(CIs) for the differences were exponentiated to provide estimates of ratio of adjusted geometric means(Test/Reference) and 90% CIs for the ratios,where FDC tablet were test and single drugs were reference.Values were back-transformed from the log scale; Test type: Superiority or Other; Ratio of adjusted geometric means = 91.63, 90% CI 2-sided [83.13 to 101.01]
Statistical Analysis 2: Comparison: RIN 150 vs Rifampicin and Isoniazid; Natural log transformed Cmax of isoniazid was analyzed using mixed effects model with sequence,period and treatment as fixed effects and participant within sequence as random effect.The adjusted mean differences and 90% CIs for the differences were exponentiated to provide estimates of ratio of adjusted geometric means(Test/Reference) and 90% CIs for the ratios,where FDC tablet were test and single drugs were reference.Values were back-transformed from the log scale; Test type: Superiority or Other; Ratio of adjusted geometric means = 107.58, 90% CI 2-sided [96.07 to 120.47]

3. Secondary Outcome: Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - ∞)]
Description: AUC (0 - ∞)= Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0 - ∞) was reported for rifampicin and isoniazid. It is obtained from AUC (0 - t) plus AUC (t - ∞).
Time Frame: as for outcome 1
Population: Pharmacokinetic parameter analysis set included all treated participants who had at least 1 estimated pharmacokinetic parameter of primary interest. Here, n=participants in the treatment group who were evaluable for this measure for specified drug of each group with reportable AUC (0 - ∞) values, respectively.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | RIN 150 | Rifampicin and Isoniazid
Number analyzed (Participants) | 27 | 27
ng*h/mL
  AUC (0 - ∞): Rifampicin (n=27, 27) | 86670 (21) | 91340 (24)
  AUC (0 - ∞): Isoniazid (n=27, 26) | 16680 (78) | 17390 (71)
Statistical Analysis 1: Comparison: RIN 150 vs Rifampicin and Isoniazid; Natural log transformed AUC(0 - ∞) of rifampicin was analyzed using mixed effects model with sequence,period and treatment as fixed effects and participant within sequence as random effect.The adjusted mean differences and 90% confidence intervals(CIs) for the differences were exponentiated to provide estimates of ratio of adjusted geometric means(Test/Reference) and 90% CIs for the ratios,where FDC tablet were test and single drugs were reference.Values were back-transformed from the log scale; Test type: Superiority or Other; Ratio of adjusted geometric means = 95.92, 90% CI 2-sided [92.54 to 99.43]
Statistical Analysis 2: Comparison: RIN 150 vs Rifampicin and Isoniazid; Natural log transformed AUC(0 - ∞) of isoniazid was analyzed using mixed effects model with sequence,period and treatment as fixed effects and participant within sequence as random effect.The adjusted mean differences and 90% confidence intervals(CIs) for the differences were exponentiated to provide estimates of ratio of adjusted geometric means(Test/Reference) and 90% CIs for the ratios,where FDC tablet were test and single drugs were reference.Values were back-transformed from the log scale; Test type: Superiority or Other; Ratio of adjusted geometric means = 102.41, 90% CI 2-sided [98.76 to 106.19]

4. Secondary Outcome: Plasma Decay Half-Life (t1/2)
Description: Plasma decay half life (t1/2) was reported for rifampicin and isoniazid.
Time Frame: as for outcome 1
Population: Pharmacokinetic parameter analysis set included all treated participants who had at least 1 estimated pharmacokinetic parameter of primary interest. Here, n=participants in the treatment group who were evaluable for this measure for specified drug of each group with reportable t½ values, respectively.
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | RIN 150 | Rifampicin and Isoniazid
Number analyzed (Participants) | 27 | 27
hour
  t1/2: Rifampicin (n=27, 27) | 3.608 (0.89531) | 3.572 (0.72948)
  t1/2: Isoniazid (n=27, 26) | 2.776 (1.4110) | 3.000 (1.4375)

5. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax)
Description: Tmax was reported for rifampicin and isoniazid.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: hour
Arm/Group | RIN 150 | Rifampicin and Isoniazid
Number analyzed (Participants) | 27 | 27
hour
  Tmax: Rifampicin | 1.67 [0.750 to 3.52] | 1.67 [0.750 to 3.52]
  Tmax: Isoniazid | 0.500 [0.250 to 2.67] | 0.500 [0.250 to 3.00]

6. Other Pre Specified Outcome: Number of Participants With Clinically Significant Changes in Vital Signs
Description: Criteria for clinical significant change in vital signs: systolic blood pressure (BP) less than (<) 90 millimeters of mercury (mmHg), diastolic BP <50 mmHg, supine and sitting heart rate <40 beats per minute (bpm) or greater than (>) 120 bpm, standing and erect heart rate <40 bpm or >140 bpm. Maximum change from baseline in systolic BP >=30 mmHg, maximum change from baseline in diastolic BP >=20 mmHg. Participants who met the criteria were reported.
Time Frame: Screening up to Day 2 of intervention period 2
Population: Safety analysis set consisted of all participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | RIN 150 | Rifampicin and Isoniazid
Number analyzed (Participants) | 27 | 27
participants | 0 | 0

7. Other Pre Specified Outcome: Number of Participants With Laboratory Test Abnormalities
Description: Criteria for laboratory tests abnormalities included: hemoglobin, hematocrit and red blood cells (less than [<] 0.8*lower limit of normal[LLN]); leucocytes (<0.6/ greater than [>] 1.5*limit of reference range [LRR]); platelets (<0.5/>1.75*LRR); neutrophils, lymphocytes (<0.8/>1.2*LRR); eosinophils, basophils, monocytes (>1.2*upper LN [ULN]); bilirubin (>1.5*ULN); aspartate aminotransferase (AST), alanine aminotransferase (ALT), alkaline phosphatase (>3*ULN); creatinine, urea (>1.3*ULN); fasting glucose (<0.6 />1.5*LRR); uric acid (>1.2*ULN); sodium (<0.95/>1.05*LRR); potassium, calcium, chloride, bicarbonate (<0.9/>1.1*LRR); albumin, total protein (<0.8/>1.2*LRR); creatine kinase (>2.0*ULN); urine red blood cells (RBCs), urine white blood cells (WBCs) (>=20 high-powered field). Total number of participants with any laboratory abnormalities was reported.
Time Frame: Screening up to Day 2 of intervention period 2
Population: Safety analysis set consisted of all participants who received at least 1 dose of study medication. Here 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure.
Measure: Number; unit: participants
Arm/Group | RIN 150 | Rifampicin and Isoniazid
Number analyzed (Participants) | 26 | 27
participants | 4 | 2

ADVERSE EVENTS:
Description: Safety analysis population included all participants who received at least 1 dose of study medication.
Arm/Group | RIN 150 | Rifampicin and Isoniazid
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/27
Other Adverse Events (participants affected / at risk) | 27/27 | 26/27
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RIN 150 (N=27) | Rifampicin and Isoniazid (N=27)
Mouth ulceration (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1
Catheter site haematoma (General disorders) | 0 | 2
Catheter site pain (General disorders) | 1 | 1
Fatigue (General disorders) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 1
Lip injury (Injury, poisoning and procedural complications) | 1 | 1
Headache (Nervous system disorders) | 1 | 1
Chromaturia (Renal and urinary disorders) | 26 | 25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.